CLINICAL TRIAL: NCT00266799
Title: A Randomized, Open-Label Trial Comparing Treatment With Either Pegylated Liposomal Doxorubicin or Capecitabine as First Line Chemotherapy for Metastatic Breast Cancer (PELICAN Trial)
Brief Title: The Efficacy and Safety of Pegylated Liposomal Doxorubicin Compared With Capecitabine as First Line Chemotherapy for Metastatic Breast Cancer (P04445/MK-2746-071)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Essex Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04445
Record Dates: First submitted 2005-12-15; First posted 2005-12-19 (Estimated); Results first posted 2011-11-16 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pegylated liposomal doxorubicin (Experimental)
  Interventions: Drug: Pegylated liposomal doxorubicin (SCH 200746)
- Capecitabine (Active Comparator)
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin (SCH 200746) — pegylated liposomal doxorubicin (50 mg/m^2 q 28 days) was administered intravenously until disease progression or unacceptable toxicity
  Arms: Pegylated liposomal doxorubicin
Drug: Capecitabine — capecitabine (1250 mg/m^2 BID x 14 days q 21 days) in tablets of 150 mg and 500 mg was administered orally, until disease progression or unacceptable toxicity
  Arms: Capecitabine

SUMMARY:
This is an open-label, multinational, randomized, multicenter trial designed to compare pegylated liposomal doxorubicin with capecitabine as first line chemotherapy of metastatic breast cancer. The primary objective of the study is to compare the time to disease progression, although overall response rates, overall survival, quality of life, time to treatment failure, and safety and tolerability will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be female.
* Patients must have metastatic disease of a cytological or histological confirmed breast cancer.
* Patients must be 18 years or older.
* Patients should have evaluable disease (at least uni-dimensionally measurable lesion according to the RECIST criteria in at least one site that has not been irradiated), however, patients who only have non-measurable/evaluable disease are not excluded. Also patients with only bone metastasis are not excluded.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) 0-2.
* Patients must have a sufficient life expectancy to be treated with chemotherapy.
* Patients must be willing and able to complete study questionnaires.
* Patients must have adequate renal function as evidenced by serum creatinine <=1.5 mg/dL, or a creatinine clearance of >=45 mL/min (if serum creatinine is > 1.5 mg/dL but <= 1.8 mg/dL).
* Patients must have adequate bone marrow function as evidenced by leukocyte count greater than 3.5 g/L, hemoglobin >=9.0 g/dL, and platelet count >=100x10^9/L.
* Patients must have adequate liver function as evidenced by bilirubin of <=1.5 times the upper limits of normal (ULN) and alkaline phosphatase <=3 times, ULN unless related to liver metastasis.
* Patients must have Sodium and Potassium values within normal limits.
* Patients whose clinical condition (co-morbidity) allows a treatment with monotherapy or who expressed their wish to be treated with monotherapy.
* Patients must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* History of receiving prior chemotherapy in the metastatic setting (Note: patients may have had

hormonal therapy or chemotherapy in the adjuvant setting; patients may have received hormonal therapy in metastatic setting, patients may have received local radiotherapy).

* Patients with positive estrogen- / progesterone-receptor status, where an endocrine therapy is indicated. However, patients progressing under hormonal therapy are not excluded.
* Patients with known hypersensitivity to doxorubicinhydrochlorid or to any of the excipients OR known hypersensitivity to capecitabine or fluorouracil or to any of the excipients.
* Patients with known DPD (dihydro pyrimidine dehydrogenase) deficiency.
* Patients who are receiving a concomitant treatment with sorivudine or its chemically related analogues, such as brivudine.
* Patients who are taking concomitant medications (except bisphosphonates) for metastatic disease, including hormonal therapy, radiation therapy, trastuzumab, or biologicals are also not permitted.
* Patients with Human epidermal growth factor receptor 2 (Her-2/neu) overexpressing tumors with the most recent evaluation as the relevant result

  * immunologically Her2neu 3+ positive
  * Her2neu-2+ positive and ´Fluorescent in-situ hybridization (FISH)´ positive
* History of treatment with capecitabine
* History of treatment with anthracyclines in the adjuvant setting exceeding cumulative doses of anthracyclines by more than 360 mg/m^2 doxorubicin (or equivalents, i.e. 600mg/m^2 epirubicine).
* Patients with anthracycline resistant disease are not permitted. Anthracycline resistance is defined as development of locally recurrent or metastatic disease while on adjuvant anthracycline therapy, or relapse less than 12 months after completion of anthracycline therapy.
* Strong remission pressure that requires polychemotherapy with the exception of patients who are not suitable for a treatment with polychemotherapy or not accepting polychemotherapy.
* Evidence of primary or metastatic malignancy involving the central nervous system unless previously treated and asymptomatic for 3 months or greater.
* Patients with reduced liver functions (evidenced by bilirubin of above 1.5 times the upper limits of normal (ULN); alkaline phosphatase above 3 times ULN (except related to liver metastasis, in which case <=5 x ULN).
* Dyspnea on exertion.
* History of cardiac disease, with New York Heart Association Class II or greater, or clinical evidence of congestive heart failure or myocardial infarct within less than six months or an left ventricular ejection fraction (LVEF) below 50%.
* Woman with childbearing potential with insufficient contraception [e.g. intra-uterine device (IUD) are regarded as sufficient] during the study period and the six months following the last study drug application. All methods based on hormonal contraception are not permitted.
* Existing pregnancy or lactation (note on pregnancy test). A negative pregnancy test for women of childbearing potential has to be in place prior randomization (Note: A pregnancy test has to be done for patients who are not postmenopausal. Postmenopausal is defined as those not having a menstrual period for 12 months in a row).
* Existing doubts on ability and willingness of the subject for cooperation.
* Participation of the subject at a clinical study within the last 30 days.
* Participation of the subject in the same clinical study at an earlier date.
* Concomitant participation in another study than the one described here.
* Abuse of drugs, alcohol, or pharmaceuticals.
* Any condition, whether medical or non-medical, that may interfere, in the opinion of the investigator, with aim of this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2006-01-13 (Actual); Primary Completion 2010-09-29 (Actual); Study Completion 2010-10-18 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 210 participants were enrolled with 105 participants randomized for treatment with PLD and 105 participants randomized for treatment with Capecitabine, of which 7 participants in the PLD group and 3 participants in the Capecitabine group were not treated.
Groups:
- Pegylated Liposomal Doxorubicin (PLD): PLD 50 mg/m^2 was administered intravenously once every 28 days. Each cycle was repeated until progress or unacceptable toxicity.
- Capecitabine: Capecitabine 1250 mg/m^2, in tablets of 150 mg and 500 mg, was administered orally twice daily (BID) for 14 consecutive days followed by a 7-day rest period. Each cycle was repeated every 21 days until progress or unacceptable toxicity.
Period: Overall Study
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) | Capecitabine
Started | 98 | 102
Completed | 62 | 68
Not Completed | 36 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) | Capecitabine | Total
Number analyzed (Participants) | 105 | 105 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] — For baseline characteristics, all 210 participants who were enrolled and randomized were incorporated , although 7 participants in the PLD group and 3 participants in the Capecitabine group were not treated.
  years | 61.4 (10.66) | 61.5 (10.59) | 61.5 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants] — For baseline characteristics, all 210 participants who were enrolled and randomized were incorporated , although 7 participants in the PLD group and 3 participants in the Capecitabine group were not treated.
  Participants
    Female | 105 | 105 | 210
    Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression (TTP) Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: TTP was defined as the time from onset of treatment with study drug until first evidence/diagnosis of progressive disease or - in the absence of any diagnosis of progressive disease - until the participant´s death. Diagnosis of progressive disease was done according to RECIST (Version 1.0) and/or investigator assessment based on RECIST. RECIST criteria used changes in the largest diameter of target/non-target lesions. Target (measurable) lesions were up to a maximum of 5 per organ & >20 mm by clinical imaging (>=10 mm with spiral CT scan). Non-target lesions were all other lesions.
Time Frame: From Day 1 (Cycle 1) until First Evidence/Diagnosis of Progressive Disease or Death
Population: Intent-to-treat (ITT): 7 in PLD group & 3 participants in Capecitabine group were missing response assessments. TTP Population: included participants in view of major protocol violations/deviations, i.e. tumor-relevant inclusion/exclusion criteria, treatment compliance, tumor assessments by RECIST with maximum 4 month interval between assessments.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) | Capecitabine
Number analyzed (Participants) | 98 | 102
Months
  By Investigator Assessment (ITT) | 6.02 [5.10 to 8.19] | 6.05 [4.27 to 9.07]
  By RECIST Criteria (ITT) | 6.58 [5.29 to 8.19] | 7.10 [4.77 to 9.53]
  By Investigator Assessment (TTP N = 63, N = 59) | 5.85 [4.37 to 7.86] | 5.88 [2.99 to 8.98]
  By RECIST Criteria (TTP N = 63, N = 59) | 6.02 [4.37 to 7.86] | 6.05 [4.08 to 9.27]
Statistical Analysis 1: Comparison: Pegylated Liposomal Doxorubicin (PLD) vs Capecitabine; By Investigator Assessment of ITT Population; Test type: Non-Inferiority or Equivalence — Non-inferiority was tested using the upper limit of the 95% CI for the hazard ratio as quantitative estimate of the minimum effect of PLD relative to capecitabine. Margin for non-inferiority was set to 1.143, reflecting an acceptable difference in TTP of 0.75 months assuming an expected median TTP of up to 6 months with the comparator. If the estimate was below margin, PLD was to be considered non-inferior to capecitabine assuming sufficient sensitivity to detect the drug effects of interest; p = 0.6686, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.76 to 1.54]
Statistical Analysis 2: Comparison: Pegylated Liposomal Doxorubicin (PLD) vs Capecitabine; By RECIST Criteria of ITT Population; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.4472, Log Rank; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.80 to 1.65]
Statistical Analysis 3: Comparison: Pegylated Liposomal Doxorubicin (PLD) vs Capecitabine; By Investigator Assessment of TTP Population; Test type: Superiority or Other; p = 0.5508, Log Rank; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.74 to 1.77]
Statistical Analysis 4: Comparison: Pegylated Liposomal Doxorubicin (PLD) vs Capecitabine; By RECIST Criteria of TTP Population; Test type: Superiority or Other; p = 0.4088, Log Rank; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.77 to 1.89]

2. Secondary Outcome: Number of Participants With an Overall Response (Complete Response [CR] + Partial Response [PR]) Between PLD and Capecitabine Treatment Groups
Description: Overall responses by investigator assessment/RECIST criteria of participant responses; CR=disappearance of target/nontarget lesions + PR=30% decrease in longest diameter sum (noting baseline sum) of target lesions. RECIST used changes in the largest diameter of target/non-target lesions. Target lesions were up to a maximum of 5 per organ & >20 mm by clinical imaging (>=10 mm with spiral CT scan). Non-target lesions were all other lesions. Evaluation of progress was repeated every 3 months (+/-7 days) post first date of lesion measurements, in detection absence until the participant´s death.
Time Frame: From Day 1 (Cycle 1) until First Evidence/Diagnosis of Progressive Disease or Death
Population: Intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: Participants
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) | Capecitabine
Number analyzed (Participants) | 105 | 105
Participants
  By Investigator Assessment - CR | 1 | 0
  By Investigator Assessment - PR | 5 | 12
  By Investigator Assessment Overall Response | 6 | 12
  By RECIST Criteria - CR | 1 | 0
  By RECIST Criteria - PR | 8 | 11
  By RECIST Criteria Overall Response | 9 | 11
Statistical Analysis 1: Comparison: Pegylated Liposomal Doxorubicin (PLD) vs Capecitabine; By Investigator Assessment; Test type: Superiority or Other; p = 0.1726, Chi-squared
Statistical Analysis 2: Comparison: Pegylated Liposomal Doxorubicin (PLD) vs Capecitabine; By RECIST Criteria; Test type: Superiority or Other; p = 0.6541, Chi-squared

3. Secondary Outcome: Overall Survival Time in the PLD and Capecitabine Treatment Groups
Description: Survival time was defined as duration time from onset of treatment with the study drug until death.
Time Frame: From Day 1 (Cycle 1) until Death
Population: ITT: 7 in PLD group and 3 participants in Capecitabine group were missing response assessments and therefore were not included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) | Capecitabine
Number analyzed (Participants) | 98 | 102
Months | 23.31 [21.44 to 27.52] | 26.79 [18.67 to 32.28]
Statistical Analysis 1: Comparison: Pegylated Liposomal Doxorubicin (PLD) vs Capecitabine; Test type: Superiority or Other; p = 0.5265, Log Rank; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.79 to 1.58]

4. Secondary Outcome: Time to Treatment Failure in the PLD and the Capecitabine Treatment Groups
Description: Time to treatment failure was defined as the duration of time from the date of the first administration of the study drug to the date of discontinuation of the study drug for any reason.
Time Frame: From Day 1 (Cycle 1) until End of Treatment
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) | Capecitabine
Number analyzed (Participants) | 98 | 102
Months | 4.60 [3.35 to 4.93] | 3.68 [2.93 to 5.85]
Statistical Analysis 1: Comparison: Pegylated Liposomal Doxorubicin (PLD) vs Capecitabine; Test type: Superiority or Other; p = 0.0841, Log Rank; p-value also given for Hazard Ratio; Hazard Ratio (HR) = 1.29

5. Secondary Outcome: Quality of Life (QoL) Measured by QoL Questionnaire (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) + Subjective Significance Questionnaire (SSQ))
Description: QoL questionnaire was an EORTC QLQ-C30 & SSQ integration. Scores on the SSQ scale ranged from 1 (very much worse) - 7 (very much better). SSQ consisted of 4 items which corresponded to core domains in the 30 Item EORTC QLQ-C30, such as improvement/deterioration in physical functioning, emotional functioning, social functioning, global QoL. Percentages were based on number of participants at each cycle & rounded to the nearest whole number. Early Withdrawal Questionnaires were obtained in 7-14 days of study drug final dose.
Time Frame: From Screening to Day 1 of every Treatment Cycle up to 12 Cycles
Population: ITT: included all randomized participants. There were only a few participants who completed more than 12 cycles due to the longer duration of each cycle.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) | Capecitabine
Number analyzed (Participants) | 105 | 105
Percentage of Participants
  Screening - Very Much Worse | 4 | 14
  Screening - Moderately Worse | 8 | 14
  Screening - A Little Worse | 12 | 24
  Screening - About the Same | 67 | 41
  Screening - A Little Better | 4 | 0
  Screening - Moderately Better | 2 | 0
  Screening - Very Much Better | 2 | 7
  Cycle 1 - Very Much Worse | 0 | 9
  Cycle 1 - Moderately Worse | 10 | 9
  Cycle 1 - A Little Worse | 22 | 9
  Cycle 1 - About the Same | 63 | 65
  Cycle 1 - A Little Better | 5 | 2
  Cycle 1 - Moderately Better | 0 | 5
  Cycle 1 - Very Much Better | 0 | 0
  Cycle 2 - Very Much Worse | 3 | 11
  Cycle 2 - Moderately Worse | 9 | 8
  Cycle 2 - A Little Worse | 25 | 15
  Cycle 2 - About the Same | 51 | 50
  Cycle 2 - A Little Better | 9 | 9
  Cycle 2 - Moderately Better | 1 | 5
  Cycle 2 - Very Much Better | 1 | 3
  Cycle 3 - Very Much Worse | 4 | 3
  Cycle 3 - Moderately Worse | 13 | 13
  Cycle 3 - A Little Worse | 13 | 23
  Cycle 3 - About the Same | 58 | 48
  Cycle 3 - A Little Better | 8 | 10
  Cycle 3 - Moderately Better | 4 | 2
  Cycle 3 - Very Much Better | 0 | 0
  Cycle 4 - Very Much Worse | 4 | 6
  Cycle 4 - Moderately Worse | 11 | 12
  Cycle 4 - A Little Worse | 26 | 22
  Cycle 4 - About the Same | 47 | 55
  Cycle 4 - A Little Better | 9 | 2
  Cycle 4 - Moderately Better | 2 | 4
  Cycle 4 - Very Much Better | 0 | 0
  Cycle 5 - Very Much Worse | 5 | 0
  Cycle 5 - Moderately Worse | 0 | 2
  Cycle 5 - A Little Worse | 21 | 19
  Cycle 5 - About the Same | 40 | 62
  Cycle 5 - A Little Better | 19 | 14
  Cycle 5 - Moderately Better | 10 | 2
  Cycle 5 - Very Much Better | 5 | 0
  Cycle 6 - Very Much Worse | 5 | 3
  Cycle 6 - Moderately Worse | 7 | 6
  Cycle 6 - A Little Worse | 9 | 11
  Cycle 6 - About the Same | 58 | 60
  Cycle 6 - A Little Better | 14 | 14
  Cycle 6 - Moderately Better | 5 | 3
  Cycle 6 - Very Much Better | 2 | 3
  Cycle 7 - Very Much Worse | 0 | 3
  Cycle 7 - Moderately Worse | 4 | 3
  Cycle 7 - A Little Worse | 17 | 23
  Cycle 7 - About the Same | 52 | 42
  Cycle 7 - A Little Better | 13 | 6
  Cycle 7 - Moderately Better | 13 | 16
  Cycle 7 - Very Much Better | 0 | 6
  Cycle 8 - Very Much Worse | 0 | 3
  Cycle 8 - Moderately Worse | 13 | 6
  Cycle 8 - A Little Worse | 17 | 16
  Cycle 8 - About the Same | 57 | 61
  Cycle 8 - A Little Better | 9 | 6
  Cycle 8 - Moderately Better | 0 | 6
  Cycle 8 - Very Much Better | 4 | 0
  Cycle 9 - Very Much Worse | 6 | 0
  Cycle 9 - Moderately Worse | 0 | 3
  Cycle 9 - A Little Worse | 25 | 21
  Cycle 9 - About the Same | 50 | 55
  Cycle 9 - A Little Better | 6 | 10
  Cycle 9 - Moderately Better | 6 | 3
  Cycle 9 - Very Much Better | 6 | 7
  Cycle 10 - Very Much Worse | 0 | 4
  Cycle 10 - Moderately Worse | 8 | 8
  Cycle 10 - A Little Worse | 17 | 13
  Cycle 10 - About the Same | 67 | 50
  Cycle 10 - A Little Better | 8 | 13
  Cycle 10 - Moderately Better | 0 | 4
  Cycle 10 - Very Much Better | 0 | 8
  Cycle 11 - Very Much Worse | 0 | 0
  Cycle 11 - Moderately Worse | 11 | 9
  Cycle 11 - A Little Worse | 0 | 13
  Cycle 11 - About the Same | 67 | 39
  Cycle 11 - A Little Better | 11 | 13
  Cycle 11 - Moderately Better | 11 | 9
  Cycle 11 - Very Much Better | 0 | 17
  Cycle 12 - Very Much Worse | 0 | 4
  Cycle 12 - Moderately Worse | 0 | 8
  Cycle 12 - A Little Worse | 11 | 13
  Cycle 12 - About the Same | 78 | 50
  Cycle 12 - A Little Better | 11 | 13
  Cycle 12 - Moderately Better | 0 | 8
  Cycle 12 - Very Much Better | 0 | 4

ADVERSE EVENTS:
Description: Due to the specification of no reason for the 2 deaths on the Capecitabine arm, these 2 events were coded as 'Death'.
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) | Capecitabine
Serious Adverse Events (participants affected / at risk) | 30/98 | 46/102
Other Adverse Events (participants affected / at risk) | 96/98 | 98/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Liposomal Doxorubicin (PLD) (N=98) | Capecitabine (N=102)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (2) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 2 (2)
ACUTE VESTIBULAR SYNDROME (Ear and labyrinth disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 2 (2)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 8 (8)
FEMORAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 2 (2)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 2 (2)
VOMITING (Gastrointestinal disorders) | 0 (0) | 2 (2)
ASTHENIA (General disorders) | 0 (0) | 1 (1)
CATHETER THROMBOSIS (General disorders) | 1 (1) | 0 (0)
CONDITION AGGRAVATED (General disorders) | 0 (0) | 1 (1)
DEATH (General disorders) | 0 (0) | 2 (2)
DISEASE PROGRESSION (General disorders) | 0 (0) | 3 (3)
FATIGUE (General disorders) | 2 (2) | 3 (4)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 4 (4) | 2 (2)
PYREXIA (General disorders) | 0 (0) | 3 (3)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 1 (2)
SUBACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (2)
HYPERSENSITIVITY (Immune system disorders) | 2 (2) | 0 (0)
CATHETER SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
FOLLICULITIS (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0)
LARYNGITIS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 1 (1)
PSEUDOMONAS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1)
WOUND INFECTION BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TRACHEAL OBSTRUCTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD POTASSIUM DECREASED (Investigations) | 0 (0) | 1 (1)
BLOOD POTASSIUM INCREASED (Investigations) | 1 (1) | 0 (0)
EAR, NOSE AND THROAT EXAMINATION ABNORMAL (Investigations) | 2 (2) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 1 (3) | 4 (4)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 (2) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 2 (2) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
CONTRALATERAL BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
METASTASES TO ABDOMINAL WALL (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO LYMPH NODES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO THORAX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
FACIAL PALSY (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 2 (2)
VERTIGO CNS ORIGIN (Nervous system disorders) | 1 (1) | 0 (0)
VITH NERVE PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 3 (3)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
BREAST PAIN (Reproductive system and breast disorders) | 1 (1) | 1 (1)
ACQUIRED TRACHEO-OESOPHAGEAL FISTULA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (7)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
THROMBOSIS (Vascular disorders) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Liposomal Doxorubicin (PLD) (N=98) | Capecitabine (N=102)
VERTIGO (Ear and labyrinth disorders) | 5 (6) | 2 (2)
LACRIMATION INCREASED (Eye disorders) | 0 (0) | 7 (7)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 11 (14)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 (5) | 9 (11)
CONSTIPATION (Gastrointestinal disorders) | 25 (43) | 10 (11)
DIARRHOEA (Gastrointestinal disorders) | 14 (18) | 42 (82)
DYSPEPSIA (Gastrointestinal disorders) | 7 (7) | 9 (13)
DYSPHAGIA (Gastrointestinal disorders) | 7 (8) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 41 (58) | 41 (57)
OESOPHAGITIS (Gastrointestinal disorders) | 5 (6) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 39 (53) | 17 (22)
VOMITING (Gastrointestinal disorders) | 18 (24) | 28 (41)
FATIGUE (General disorders) | 53 (81) | 54 (89)
OEDEMA PERIPHERAL (General disorders) | 7 (7) | 12 (12)
PYREXIA (General disorders) | 5 (5) | 6 (9)
HYPERSENSITIVITY (Immune system disorders) | 10 (12) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 4 (5) | 8 (11)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 10 (12) | 15 (23)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 11 (14) | 12 (22)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 8 (10) | 6 (9)
BLOOD BILIRUBIN INCREASED (Investigations) | 2 (3) | 13 (38)
BLOOD CREATININE INCREASED (Investigations) | 3 (3) | 8 (11)
EAR, NOSE AND THROAT EXAMINATION ABNORMAL (Investigations) | 42 (57) | 17 (21)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 8 (11) | 2 (2)
HAEMOGLOBIN DECREASED (Investigations) | 25 (50) | 19 (41)
NEUTROPHIL COUNT DECREASED (Investigations) | 18 (55) | 9 (20)
PLATELET COUNT DECREASED (Investigations) | 6 (10) | 7 (12)
WEIGHT DECREASED (Investigations) | 5 (7) | 7 (8)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 37 (106) | 16 (37)
ANOREXIA (Metabolism and nutrition disorders) | 12 (13) | 15 (18)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 13 (18) | 10 (10)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 9 (13) | 15 (18)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 (11) | 3 (12)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (8) | 2 (4)
DIZZINESS (Nervous system disorders) | 3 (3) | 10 (15)
DYSGEUSIA (Nervous system disorders) | 2 (2) | 8 (10)
HEADACHE (Nervous system disorders) | 6 (6) | 5 (5)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 17 (23) | 25 (29)
DEPRESSION (Psychiatric disorders) | 2 (2) | 8 (9)
INSOMNIA (Psychiatric disorders) | 9 (10) | 7 (9)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 11 (12)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 14 (19) | 22 (26)
ALOPECIA (Skin and subcutaneous tissue disorders) | 27 (27) | 10 (11)
DRY SKIN (Skin and subcutaneous tissue disorders) | 10 (11) | 6 (6)
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 7 (8) | 7 (8)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 8 (12) | 3 (4)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 9 (12) | 12 (16)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 65 (227) | 68 (248)
PRURITUS (Skin and subcutaneous tissue disorders) | 8 (11) | 2 (2)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 6 (9) | 3 (3)
FLUSHING (Vascular disorders) | 6 (7) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If investigator wishes to publish study information, a copy of the manuscript must be provided to sponsor for review at least 60 days before submission of publication/presentation. In the event issues arise regarding scientific integrity/regulatory compliance, sponsor will review these issues with investigator. Investigator will not publish data derived from the individual site until 12 months after conclusion/abandonment/termination of study at all sites.